CLINICAL TRIAL: NCT05987488
Title: Early Clinical Development of a Live, Attenuated Combination Vaccine Against Shigella and ETEC Diarrhoea: Phase 1b Clinical Trial of ShigETEC Vaccine in Bangladeshi Adults and Three Paediatric Age Groups
Brief Title: ShigETEC Vaccine Study in Bangladesh
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eveliqure Biotechnologies GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PR-19067
Record Dates: First submitted 2023-07-25; First posted 2023-08-14 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers
Keywords: Shigella; Enterotoxigenic Escherichia Coli
MeSH Terms: conditions — Dysentery, Bacillary | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ShigETEC vaccine (Experimental): The vaccine will consist of a suspension of a live, attenuated Shigella bacterial strain (a clinical isolate of Shigella flexneri 2457T strain) into which the genes for nontoxic forms of the ETEC heatlabile toxin B subunit (LTB) and a mutant heat stable toxin (STm) have been inserted.
  Interventions: Biological: ShigETEC live, attenuated, oral vaccine
- Placebo (Placebo Comparator): A saline solution with corn starch
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ShigETEC live, attenuated, oral vaccine — Vaccine will be delivered orally.
  Stage 1:
  Adults (18-45 years) will intake the vaccine 3 times 14 days apart in a dose escalating setting with two different doses.
  Stage 2:
  Children (2-5 years), Toddlers(12-23 months), Younger children (6-11 months) will intake the vaccine 3 times 14 days apart in a dose escalating setting with three different doses.
  Arms: ShigETEC vaccine
Other: Placebo — Placebo will be delivered orally.
  Stage 1:
  Adults (18-45 years) will intake the placebo 3 times 14 days apart
  Stage 2:
  Children (2-5 years), Toddlers(12-23 months), Younger children (6-11 months) will intake the placebo 3 times 14 days apart.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test ShigETEC vaccine, a combination vaccine against Shigella and ETEC diarrhoea in Bangladeshi adults (aged 18-45 years) and paediatric participants of three different age groups (aged 2-5 years, 12-23 months and 6-11 months).

The main question[s] it aims to answer are:

* Safety and clinical tolerability of the vaccine
* Immune responses generated by the vaccine In the age-descending dose-escalating study
* Adult participants will be divided into 2 escalating dose cohorts
* Each age group of paediatric participants will be divided into 3 escalating dose cohorts
* Participants in each cohort will receive three doses of vaccine/placebo two weeks apart
* Solicited and unsolicited adverse events (AE) and serious adverse events (SAE) will be monitored after each vaccination dose
* Stool samples will be collected for immunological analysis and shedding of vaccine strain
* Blood samples will be collected for immunological analysis

DETAILED DESCRIPTION:
A double-blind, randomized, placebo-controlled, age-descending and dose-escalating phase 1b clinical trial will be carried out in Bangladeshi adults and three paediatric age groups to evaluate the safety, clinical tolerance, and immunogenicity of ShigETEC, a live, attenuated Shigella/ETEC combination vaccine.

Objectives of the study

Primary Objectives:

To evaluate the safety and clinical tolerability of oral ShigETEC vaccine in Bangladeshi adults and different age groups of paediatric participants by monitoring the occurrence and severity of clinical signs and symptoms after administration of each of the three vaccinations.

Secondary Objectives:

* To evaluate the immune response to Shigella and ETEC (Enterotoxigenic Escherichia coli) antigens in blood and stool following administration of ShigETEC vaccine.
* To assess the fecal shedding of ShigETEC following ingestion.

The age-descending study will start testing the vaccine in healthy adults (aged 18-45 years) and move subsequently into three different paediatric age groups (aged 2-5 years, 12-23 months and 6-11 months). In the adult participants (group A), fifty-four participants will be enrolled and divided into 3 escalating dose cohorts. Each cohort of 18 healthy adults (12 vaccinees and 6 placebo recipients) will be randomized to receive three times vaccine/placebo two weeks apart. The first adult cohort (cohort A1) will receive the optimal vaccine dose (OVD) found in Phase I Europe trial (5x10^10 CFU). Cohort A2 will be given 4-fold higher dose than cohort A1 (2x10^11 CFU). Cohort A3 will receive a lower dose according to DSMB decision (2x10^9 CFU).

In each of the 2-5 years (group B), 12-23 months (group C), and 6-11 months age group (group D), 48 participants will be enrolled and divided into 3 escalating dose cohorts with 16 participants in each cohort (12 vaccinees and 4 placebo recipients). B1 cohort will be immunized with 25-fold lower than the OVD in EU (Europe) Phase 1 trial (2x10^9CFU). Cohorts B2 and B3 will be given higher doses in 5-fold increments, and thus cohort B2 will receive 1x10^10 CFU and cohort B3 will receive the OVD in EU Phase 1 trial (5x10^10 CFU). Cohort C1 will be vaccinated with 25-fold lower than the OVD in group B. Cohorts C2 and C3 will receive higher doses in 5-fold increments. Cohort D1 will be given 25- fold lower than the OVD in group C. Cohorts D2 and D3 will receive higher doses in 5-fold increments.

Recruitment, screening, and consenting of the participants will take place at the urban field site of icddr,b in Mirpur. In each cohort, the first dose and immediate safety evaluation will be conducted at the Clinical Trial Unit (CTU), an inpatient facility, where the participants will be closely monitored for 24 hours post-vaccination. If the initial dose is deemed safe, all participants will return to the CTU to receive the second and third time vaccine or placebo on an outpatient basis. Follow-up visits will take place 7 days after each dosing and 28 days after last dosing at the Mirpur field office.

Primary safety endpoint:

1. Solicited reactogenicity
2. Unsolicited adverse event (AE)
3. Serious adverse event (SAE)

Secondary immunogenicity endpoints:

1. Changes of antibody responses to antigens from baseline to each visit after vaccination:

   * Antibody responses IgG (Immunglobulin G) and IgA (Immunglobulin A) in all age groups in serum
   * IgA in lymphocyte supernatant (ALS) and fecal extract
2. Functional antibodies:

   * ETEC toxins neutralization titers
   * Serum bactericidal activity
   * Inhibition of bacterial adherence and entry to human colon epithelial cells
3. Antibody responses to Shigella and ETEC proteins and peptides
4. Antibody avidity against LT, ST and selected Shigella antigens

Secondary shedding endpoint:

Intestinal replication of the ShigETEC vaccine

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults, children, toddlers, and infants aged between 18-45 years, 2-5 years, 12-23 months, and 6-11 months, respectively at the time of vaccination.
* Free of obvious health problems as determined by medical history and clinical examination before entering into the study.
* Normal bowel habits.
* Informed consent form signed.
* Negative pregnancy tests before each vaccination for females of childbearing potential. Adult participants agree to use birth control steps or abstinence.

Exclusion Criteria:

* Nursing and breast-feeding women.
* Presence of any known significant medical or psychiatric condition / systemic disorder.
* History of congenital abdominal disorders, intussusception, abdominal surgery, any other congenital disorder, any neurologic disorders or seizures.
* Clinically significant abnormalities in screening hematology, serum chemistry.
* Known or suspected HIV, hepatitis infection.
* Clinical evidence of active gastrointestinal illness or acute disease at the time of enrolment.
* Prior receipt of any Shigella or ETEC vaccine, blood transfusion or blood products.
* History of febrile illness within 48 hours prior to vaccination or fever at the time of immunization.
* History of diarrhoea within 7 days and / or acute diarrhoea due to culture confirmed Shigella or ETEC infections within one month prior to vaccination.
* Screening stool positive for any Shigella or ETEC strain by culture.
* Participation in research involving another investigational product within 30 days before before planned date of first vaccination concurrent participation in another clinical trial.
* Receipt of antimicrobial drugs for any reason within 7 days before vaccination.
* Allergy to quinolone, sulfa, and penicillin classes of antibiotics
* Any conditions which, in the opinion of the investigator, might jeopardize the safety of study participants or interfere with the evaluation of the study objectives.

Ages: 6 Months to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 196 (Actual)
Dates: Start 2023-11-26 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Reactogenicity | 72 hours after vaccination
  Solicited adverse events in participants after vaccination. ShigETEC vaccine may result in symptoms similar to infection with Shigella or ETEC including fever, decreased appetite, irritability, decreased activity, abdominal pain, nausea, vomiting, loose stool, diarrhoea, dysentery, bloating, excess flatulence and constipation.
Unsolicited adverse event (AE) | From first vaccination throughout 56 days
  Any untoward medical occurrence in study participants during the conduct of a clinical trial, for which there is no or less possibility that the drug caused the event.
Serious adverse event (SAE) | From first vaccination throughout 56 days
  Adverse event(s) classified as serious per definition.

SECONDARY OUTCOMES:
Antigen-specific Antibody titers induced by ShigETEC | From the day of first vaccination throughout 56 days in a 14 day interval
  Changes in IgG and IgA in plasma/serum, IgA in ALS and fecal extract to specific antigens from baseline to each visit after vaccination.
Functional antibodies induced by ShigETEC- neutralization | From the day of first vaccination throughout 56 days in a 14 day interval
  ETEC toxins neutralization titers
  * Serum bactericidal activity
  * Inhibition of bacterial adherence and entry to human colon epithelial cells
Characterization of the antibody repertoire induced by ShigETEC | From the day of first vaccination throughout 56 days in a 14 day interval
  Mapping of the vaccine-induced antibody for the entire Shigella proteome and ETEC toxin by high-resolution peptide and protein microarray assay.
Antibody avidity induced by ShigETEC | From the day of first vaccination throughout 56 days in a 14 day interval
  Antigen-antibody binding avidity
Shedding of vaccine in stool | From the day of first vaccination throughout 56 days
  Assessment of intestinal replication of the ShigETEC vaccine
Functional antibodies induced by ShigETEC - SBA | From the day of first vaccination throughout 56 days in a 14 day interval
  Serum bactericidal activity
Functional antibodies induced by ShigETEC - adherence | From the day of first vaccination throughout 56 days in a 14 day interval
  Inhibition of bacterial adherence and entry to human colon epithelial cells

CONTACTS AND LOCATIONS:
Locations (1):
- International Centre for Diarrhoeal Diseases Research, Bangladesh (icddr,b), Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No